CLINICAL TRIAL: NCT00207818
Title: Treatment of Cutaneous Ulcers With a Novel Biological Dressing
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LOEX 005; 29478 Health Canada
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Venous Ulcers
Keywords: tissue engineered wound dressing; autologous skin substitute; biological dressing; wound care
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: self assembled skin substitute (SASS) — Wound care with self assembled skin substitute (SASS)

SUMMARY:
The aim of the study is to evaluate the effect of a biological dressing on the healing process of venous ulcers. The dressing is a reconstructed skin substitute made with the patients own cells.

DETAILED DESCRIPTION:
The hypothesis of this trial is that the cutaneous model SASS, a dermal epidermal skin substitute, created by the LOEX could be as high-performant, or even better, than the one's already existent in North America for the wound care. We anticipate showing on 6 patients that ulcer that did not close with conventional treatment, will heal or at least improve with this treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women from 18 to 85 years old
2. Have a venous ulcer or a mixed ulcer

Exclusion Criteria:

Diabetes Mental deficiency Hepatitis holder (A-B-C) HIV positive Pregnancy or lactation Corticosteroids therapy Radiotherapy Chemotherapy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 1999-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
wound closure

SECONDARY OUTCOMES:
% of healing at 6 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Francois A Auger, MD, Principal Investigator — Centre hospitalier affilié universitaire de Québec; Lucie Germain, Ph.D., Study Director — Centre hospitalier affilié universitaire de Québec
Locations (1):
- Centre hospitalier affilie universitaire de Quebec, Québec, Quebec, Canada

REFERENCES:
- [Background] Pouliot R, Larouche D, Auger FA, Juhasz J, Xu W, Li H, Germain L. Reconstructed human skin produced in vitro and grafted on athymic mice. Transplantation. 2002 Jun 15;73(11):1751-7. doi: 10.1097/00007890-200206150-00010. PMID 12084997
- [Background] Michel M, L'Heureux N, Pouliot R, Xu W, Auger FA, Germain L. Characterization of a new tissue-engineered human skin equivalent with hair. In Vitro Cell Dev Biol Anim. 1999 Jun;35(6):318-26. doi: 10.1007/s11626-999-0081-x. PMID 10476918
- See also: LOEX research laboratory website — http://www.loex.qc.ca